CLINICAL TRIAL: NCT05570773
Title: Effects of Peer Support and Progressive Relaxation Exercises on Sleep Quality and Anxiety in Midwifery Students During COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: Effects of Peer Support and Progressive Relaxation Exercises on Sleep Quality and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Elif DAĞLI, Lecturer Doctor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Relaxation
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Anxiety; Sleep Disturbance
MeSH Terms: conditions — Anxiety Disorders; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- peer support program (Experimental): A researcher and peer tutors met students in an online session for 30 minutes every day between 21:00 and 21:30 before bedtime for 30 days. These sessions focused on academic problem solving and academic encouragement of students. In addition, peer tutors and students shared their contact information and continued their sharing by talking on the phone and messaging in the chat group 24/7.
  Selection and education of peer tutors: 5 peers with strong communication skills and high academic achievement were selected among the 4th-year volunteer students. These 5 volunteers were selected among students who were not included in the sample, had an appropriate level of anxiety (anxiety score ≤36), and had good sleep quality (PSQI score ≤5). A theoretical and practical session was held with them. In these sessions, peer-supported education was explained and necessary information was given about its purpose and how it was performed.
  Interventions: Other: peer support program
- progressive relaxation exercise group (Experimental): The importance of the exercise and how it should be done were explained by the researcher Mixed teaching methods, including lecturing, demonstration, question-answer, and discussion were, used as education methods. The sessions were carried out online by a researcher who is an expert in the field of PRE for 30 minutes every day between 21:00 and 21:30 before bedtime for 30 days.
  Interventions: Other: peer support program
- control group (No Intervention): The students who formed the control group through randomization were given information about the research, and then they submitted informed consent. Control group students were given the same questionnaire as a pre-and-post-test applied in the intervention groups, but no intervention was applied.

INTERVENTIONS:
Other: peer support program — Peer support: It has been suggested that peer support provides an alternative way for students to learn and makes a positive contribution to both academic and psychosocial aspects of higher education (Hogan, Fox, Barratt-See 2017). Peer academic support involves academic encouragement (support for lowering exam-related stress and motivation for lessons) and solving students' academic problems (answering questions about lessons, sharing study habits, studying together, answering questions about assignments)
  Other Names: progressive relaxation exercises program
  Arms: peer support program; progressive relaxation exercise group

SUMMARY:
The effect of peer support and progressive relaxation exercise programs on midwifery students' sleep and anxiety levels in the COVID-19 pandemic was investigated in the present research. One hundred and four subjects were found eligible for the study according to the inclusion criteria, and they were grouped into three: the peer support program group (PSP) (n=34), the progressive relaxation exercise group (PRE) (n=35), and control group (n=35). The PRE group was given an online relaxation exercise program. The PSP group was given an online peer support program. The data collection tools included a descriptive data form, State-Trait Anxiety Inventory (STAI-I-II), and Pittsburgh Sleep Quality Index (PSQI). The scores of the groups that they obtained from the pre-test application of the STAI-I and PSQI did not yield a statistically significant difference. The scores that PRE and PSP groups obtained from the post-test application of the STAI-I and PSQI were lower than the score that was obtained by the control group on the post-test application of the measures, and difference was evaluated to be significant. Although the mechanisms of action of these two methods are different, it has been observed that they have similar effects in improving anxiety levels and sleep quality.

DETAILED DESCRIPTION:
This is a randomized, controlled intervention trial. It was carried out according to CONSORT guidelines between February 12 and March 28, 2021 with students who were studying midwifery at a state university.

Randomization Three hundred and sixty students from the midwifery department made up the population of the study, and the sample consisted of three hundred and thirteen students that agreed to join the study. We excluded some subjects from the study according to the exclusion criteria. The remaining one hundred and forty-four subjects were randomly divided into groups as PRE, PSP, and controls through randomization by assigning consecutive numbers to them via computer software (https://www.randomizer.org/). Accordingly, forty-eight students were assigned to the PRE group, forty-eight to the PSP group, and forty-eight to the control group. After the randomization step, 8 students from the PRE group, 10 from the PSP group, and 12 from the control group, who did not want to continue, were excluded from the study. During the follow-up period, 3 students from the PRE group and 2 students from the PSP group were excluded because they did not achieve 80% attendance. Since five subjects (two, PRE group; two, PSP group; one, control group) were unavailable during the data analysis stage, their final measurements could not be made, and therefore they were excluded. The study was completed with a total of 104 students, including 35 in the PRE group, 34 in the PSP group, and 35 in the control group. First, all 3 groups filled out the questionnaires as a pre-test application. At the end of 30 days, the groups filled out the questionnaires as a post-test. It took approximately 10-15 minutes to fill out the questionnaires.

Intervention groups PRE group The importance of the exercise and how it should be done were explained by the researcher Mixed teaching methods, including lecturing, demonstration, question-answer, and discussion were, used as education methods. The sessions were carried out online by a researcher who is an expert in the field of PRE for 30 minutes every day between 21:00 and 21:30 before bedtime for 30 days.

Steps of progressive relaxation exercises: This progressive relaxation technique developed by Jacobson is one of the easiest to learn and practice. PRE is a holistic approach based on the controlled, voluntary, regular, and successive active contraction and passive relaxation of major muscle groups. The person is asked to wear comfortable clothes, relax as much as possible, and breathe slowly and deeply. This technique, which can be applied sitting or lying down, can also be performed with music to contribute to the relaxation of the individual.

The education begins with diaphragmatic breathing exercises and continues with PRE. In this exercise, the patient positions one of his/her hand on his/her chest and the other on the mid-abdomen, and then told to breathe in slowly and deeply through the nose, counting to 4, hold the air counting to 4 again, and exhale by pursing lips while exhaling. In diaphragmatic breathing, the abdomen is expected to be inflated as much as possible while breathing in through the nose. While performing the exercise, the sensory, visual, and tactile stimuli given to the patient are gradually reduced and made difficult. The exercise is repeated 2-3 times, and then the patient is allowed to rest between the sessions.

PRE is applied from the bottom to the top, starting from the feet to the lower extremity, trunk, upper extremity, and facial muscles, respectively. The person is asked to relax and start by giving their attention to their feet when they are ready, and focus on their feet for a while and perceive how they feel. The person is told to take a deep breath and slowly tighten their foot for 10-20 seconds, and then release the foot muscles while exhaling and feel the loose and flexible state of the foot for 30-40 seconds. During relaxation, deep, slow breathing is continued while moving the upper part of the body. A total of 15 zones/muscle groups are exercised with one repetition, without giving a break. After each contraction and relaxation process, slow and deep diaphragmatic breathing exercises should be performed several times before moving on to a new muscle group. After all the muscles are contracted and released in turn, now, all the muscles are contracted simultaneously while breathing in and are simultaneously released again while exhaling. Then, the exercises are completed with slow and deep diaphragmatic breathing.

PSP group A researcher and peer tutors met students in an online session for 30 minutes every day between 21:00 and 21:30 before bedtime for 30 days. These sessions focused on academic problem solving and academic encouragement of students. In addition, peer tutors and students shared their contact information and continued their sharing by talking on the phone and messaging in the chat group 24/7.

Selection and education of peer tutors: 5 peers with strong communication skills and high academic achievement were selected among the 4th-year volunteer students. These 5 volunteers were selected among students who were not included in the sample, had an appropriate level of anxiety (anxiety score ≤36), and had good sleep quality (PSQI score ≤5). A theoretical and practical session was held with them. In these sessions, peer-supported education was explained and necessary information was given about its purpose and how it was performed.

Peer support: It has been suggested that peer support provides an alternative way for students to learn and makes a positive contribution to both academic and psychosocial aspects of higher education. Peer academic support involves academic encouragement (support for lowering exam-related stress and motivation for lessons) and solving students' academic problems (answering questions about lessons, sharing study habits, studying together, answering questions about assignments).

Control group The students who formed the control group through randomization were given information about the research, and then they submitted informed consent. Control group students were given the same questionnaire as a pre-and-post-test applied in the intervention groups, but no intervention was applied.

Data collection Data collection tools included the State and Trait Anxiety Inventory, which was developed by Spielberger, (STAI-I-II), the Pittsburgh Sleep Quality Index (PSQI), and a descriptive information form designed to collect socio-demographic information.

ELIGIBILITY:
Inclusion Criteria:

* did not have sleep apnea,
* did not musculoskeletal disease
* did not cardio-pulmonary disease
* did not psychiatric disease
* did not use drugs, cigarettes, alcohol
* SAI score of >36 (anxiety)
* PSQI score of >5 (poor sleep quality)

Exclusion Criteria:

* Clinical diagnosis of sleep apnea
* musculoskeletal disease
* cardio-pulmonary disease
* psychiatric disease
* history of drugs, smoking, and alcohol
* SAI score of ≤36 (no anxiety),
* PSQI score of ≤5 (good sleep quality)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
State and Trait Anxiety Inventory | 16 weeks
  questionnaire

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 16 weeks
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fatma TOPKARA, Dr., Study Chair — Eskişehir Osmangazi University
Locations (1):
- Cukurova University, Adana, Balcalı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No